CLINICAL TRIAL: NCT02702986
Title: Immunostimulating Interstitial Laser Thermotherapy in Patients With Locally Advanced Pancreatic Cancer: Results of a Prospective, Open, Non Comparative Study
Brief Title: Safety and Feasibility of imILT Locally Advanced Pancreatic Cancer (LAPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Principal Investigator, Salvatore Paiella, MD, MD, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2015-001
Record Dates: First submitted 2016-02-14; First posted 2016-03-09 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imILT of pancreatic cancer (Experimental): 10 patients suffering from LAPC will be submitted to immunostimulating interstitial laser thermotherapy (imILT) in a single-arm setting
  Interventions: Procedure: immunostimulating Interstitial Laser Thermotherapy; Device: Laser

INTERVENTIONS:
Procedure: immunostimulating Interstitial Laser Thermotherapy — Through a laparotomy a laser device will be inserted into the locally advanced pancreatic cancer.
  Other Names: imILT
Device: Laser

SUMMARY:
10 Patients with Locally Advanced Pancreatic Cancer, no further responsive to neoadjuvant treatments but with a Stage-III disease will be submitted to imILT (Immunostimulating Interstitial Laser Thermotherapy). Safety and feasibility of imILT on LAPC will be evaluated as primary objective. Secondary objectives will be QoL after imILT, study of the immune reaction after imILT, oncological analysis of patients suffering from LAPC submitted to imILT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III locally advanced pancreatic cancer
* No further neoadjuvant treatments are doable
* Eastern Cooperative Oncology Group performance status < 1

Exclusion Criteria:

* No other concomitant oncological treatments (hormonal, immunotherapies, etc)
* Suffering from other neoplasms
* Suffering from HIV
* Suffering from autoimmune diseases
* Concomitant medication with steroids

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 24 months

SECONDARY OUTCOMES:
The immunostimulating effects of imILT | Up to 24 months
  This will be determined by measuring plasma levels of various pro and anti-inflammatory cytokines and immune-related cells
Overall Survival | Up to 24 months
Progression free survival (PFS) | Up to 24 months
Disease specific survival (DSS) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona Hospital, Verona, Italy

REFERENCES:
- [Result] Haraldsdottir KH, Ivarsson K, Jansner K, Stenram U, Tranberg KG. Changes in immunocompetent cells after interstitial laser thermotherapy of breast cancer. Cancer Immunol Immunother. 2011 Jun;60(6):847-56. doi: 10.1007/s00262-011-0992-8. Epub 2011 Mar 13. PMID 21400025
- [Result] Ivarsson K, Myllymaki L, Jansner K, Stenram U, Tranberg KG. Resistance to tumour challenge after tumour laser thermotherapy is associated with a cellular immune response. Br J Cancer. 2005 Aug 22;93(4):435-40. doi: 10.1038/sj.bjc.6602718. PMID 16091763
- [Result] Tranberg KG, Moller PH, Hannesson P, Stenram U. Interstitial laser treatment of malignant tumours: initial experience. Eur J Surg Oncol. 1996 Feb;22(1):47-54. doi: 10.1016/s0748-7983(96)91451-1. PMID 8846867
- [Result] Tranberg KG, Myllymaki L, Moller PH, Ivarsson K, Sjogren HO, Stenram U. Interstitial laser thermotherapy of a rat liver adenocarcinoma. J Xray Sci Technol. 2002 Jan 1;10(3):177-85. PMID 22388047
- [Result] Ivarsson K, Myllymaki L, Jansner K, Bruun A, Stenram U, Tranberg KG. Heat shock protein 70 (HSP70) after laser thermotherapy of an adenocarcinoma transplanted into rat liver. Anticancer Res. 2003 Sep-Oct;23(5A):3703-12. PMID 14666667
- [Derived] Paiella S, Casetti L, Ewald J, Marchese U, D'Onofrio M, Garnier J, Landoni L, Gilabert M, Manzini G, Esposito A, Secchettin E, Malleo G, Lionetto G, De Pastena M, Bassi C, Delpero JR, Salvia R, Turrini O. Laser Treatment of Pancreatic Cancer with Immunostimulating Interstitial Laser Thermotherapy Protocol: Safety and Feasibility Results From Two Phase 2a Studies. J Surg Res. 2021 Mar;259:1-7. doi: 10.1016/j.jss.2020.10.027. Epub 2020 Dec 2. PMID 33278792